CLINICAL TRIAL: NCT04596163
Title: Transversus Thoracis Muscle Plane Block for Acute and Chronic Pain Management in Cardiac Surgical Patients Requiring Sternotomy: a Prospective Randomized Controlled Trial
Brief Title: Transversus Thoracis Muscle Plane Block for Sternotomy Pain in Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, WONG MAN KIN, Honorary Clinical Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020.371-T
Record Dates: First submitted 2020-10-06; First posted 2020-10-22 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Pain, Postoperative; Surgical Wound; Cardiac Event
Keywords: Regional anaesthesia; Cardiac surgery
MeSH Terms: conditions — Pain, Postoperative; Surgical Wound; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Single-centred, double-blinded, randomized, placebo-controlled trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Ultrasound guided Regional block using 0.25% levobupivacaine (local anaesthetic agent) 20ml (50mg) on each side of the sternum over 1-2 minutes after general anaesthesia before surgery.
  Interventions: Procedure: Transversus thoracis muscle plane block
- Control (Placebo Comparator): Ultrasound guided Regional block using 20ml of 0.9% normal saline on each side of the sternum after general anaesthesia before surgery.
  Interventions: Procedure: Transversus thoracis muscle plane block

INTERVENTIONS:
Procedure: Transversus thoracis muscle plane block — After general anaesthesia, transversus thoracis plane (TTP) block, a kind of regional block will be performed near both sides of the sternum under ultrasound guidance using either levobupivacaine or normal saline to both groups of patients. The end point for injection is the fluid spread along the plane just superficial to the transversus thoracis muscle, together with the downward displacement of the pleura.

SUMMARY:
Sternotomy pain is usually significant after cardiac surgery. Analgesic options for sternotomy in cardiac surgery are often limited. Poorly controlled acute pain is an important factor to development of chronic postsurgical pain. The transversus thoracis muscle plane (TTP) block is a novel technique that provides analgesia to anterior chest wall. A double-blinded RCT is conducted to assess the efficacy of applying TTP block as an adjunct to analgesia in cardiac surgery.

DETAILED DESCRIPTION:
Chronic postsurgical pain (CPSP) is defined as the persistence of pain at surgical site or referred area, at least 3 months following the surgical procedure. CPSP after median sternotomy is not uncommon after cardiac surgery. The reported incidence ranges from 28% to 56% up to 2 years postoperatively. A number of factors can contribute to the variation in incidence, including the variations in presentation of chronic post-sternotomy pain and under-reporting from patients. Given the nature of cardiac surgery and considerable anxiety of patients at perioperative period, patients would tend to live with the chronic pain and rationalize it as a normal consequence of the surgery. Patients therefore may not report any symptoms, resulting in a delay in diagnosis of chronic post-sternotomy pain.

The mechanisms for development of CPSP after sternotomy are not fully known. The up-regulation, activation and neural sensitization during the acute pain phase are important factors to the development of chronic pain. Causes of pain from sternotomy include neuropathy from anterior intercostal nerves entrapment or injury during surgical dissection and internal mammary artery harvesting, musculoskeletal injury from surgical incision and dissection, sternal fracture or incomplete bone healing, and development of sternal wound infections. Poorly controlled acute pain in the perioperative period can trigger central sensitization, a stepwise modification of spinal pain pathways involving protein synthesis and synaptic strength, which can lead to hyperalgesia and chronic pain. Therefore, good perioperative acute pain control not only provides postoperative pain relief, but also prevents occurrence of chronic pain.

In most centres, opioids such as fentanyl and morphine are used mainly for the management of acute pain after cardiac surgery. However, perioperative opioids are known to be associated with dose-dependent side effects such as nausea and vomiting, pruritis, respiratory depression, postoperative chronic opioid use and increased risk of chronic pain. Multimodal approach such as the use of NSAIDs may not be optimal after cardiac surgery due to the risk of bleeding and renal failure. Regional analgesia has opioid-sparing effect and seems to be a good choice for perioperative anaglesia. Regional techniques such as thoracic epidural and paravertebral blocks have been described but they are not ideal due to the potential complications from systemic heparinization in cardiac surgery. Erector spinae plane (ESP) block was reported to decrease perioperative morphine consumption and early postoperative pain score. However, the transverse process tip is not always easy to visualize on ultrasound, especially in obese patients, resulting in variation in ESP block efficacy.

Transversus thoracis muscle plane (TTP) block covers the anterior branches of intercostal nerves T2 to T6. It has been described in cardiac surgical patients that provides analgesia for sternotomy. TTP block is a superficial block and therefore is relatively safe when compared with thoracic epidural and paravertebral nerve block during heparinization. The investigators hypothesized that pre-emptive TTP block can provide effective perioperative analgesia and prevent the occurrence of CPSP in cardiac surgical patients requiring median sternotomy. A prospective, double-blinded randomized controlled trial was conducted to assess the analgesic efficacy of TTP block in open cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Elective CABG, aortic valve repair/replacement, mitral valve repair/replacement, or combined CABG/valve procedure

Exclusion Criteria:

* emergency surgery
* redo surgery
* history of thoracotomy or mastectomy
* history of chronic pain or regular analgesic use (except paracetamol and NSAID)
* history of psychiatric illnesses or illicit drug use
* renal failure with eGFR <30ml/min or on renal replacement therapy
* mortality or require re-sternotomy within 24h after operation
* intraoperative use of remifentanil
* unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2022-10-22 (Actual); Study Completion 2023-04-22 (Actual)

PRIMARY OUTCOMES:
Opioid consumption | Once at the end of the surgery
  The total amount of opioid (mg) used during the surgery

SECONDARY OUTCOMES:
Percentage blood pressure change | From 5 minutes before skin incision to 10 minutes after skin incision at 1 minute interval ( a total of 15 time point)
  The percentage changes in systolic blood pressure (SBP), diastolic blood pressure (DBP), mean arterial pressure (MAP) between the baseline (before surgery) and within 10 minutes after skin incision for sternotomy
Percentage heart rate change | From 5 minutes before incision to 10 minutes after skin incision at 1 minute interval (a total of 15 time points)
  Heart rate (HR) between the baseline (before surgery) and their peaks within 10 minutes of skin incision for sternotomy.
Morphine consumption | up to 72 hours postoperatively
  The amount of morphine (mg) used after the surgery for pain control
Length of hospital stay | Immediately after the surgery up to the day of patient discharge
  duration of hospital stay (in days)
Intensive Care unit (ICU) stay | Immediately after the surgery up to the time of ICU discharge
  duration of ICU stay (in hours)
Pain score | At 8, 12, 24, 48 and 72 hours after TTP block and on day 7 after surgery (6 time points).
  A visual analogue scale of 0-10 (0=no pain, 10=worst pain) will be used to grade the pain score. Patients will be asked to rate the intensity of postoperative pain at rest and on three maximal coughs.
Peak expiratory flow rate | Once as baseline on the day before operation and at 6 time points after surgery (ie. at 8, 12, 24, 48, 72 hours after block and on day 7 after surgery).
  Measured with a spirometer at baseline on the day before operation and postoperatively at the time of assessing pain score. The higher the result means the better the lung function of the patient.
Forced expiratory volume in 1 second | Once as baseline on the day before operation and at 6 time points after surgery (ie. at 8, 12, 24, 48, 72 hours after block and on day 7 after surgery).
  Measured with a spirometer at baseline on the day before operation and postoperatively at the time of assessing pain score. The higher the result means the better the lung function of the patient.
Brief Pain Interference Scale | at 3-month and 6-month after surgery
  It will be used to evaluate the extent of pain interfering with various components of functioning, including physical functioning, emotional functioning and sleep within the last 24 hours at 3 and 6 months after surgery (a score of 0-10; 0=no interference at all, 10= the worst interference due to pain).
Pain Catastrophizing Scale | at 3-month and 6-month after surgery
  Pain Catastrophizing Scale (HK-PCS) will be used to assess patients' negative cognitive-affective responses to pain within the last 24 hours at 3 and 6 months after surgery. Score 0-100 (0=no pain related anxiety; 100=most severe pain related anxiety)

CONTACTS AND LOCATIONS:
Overall Officials: Henry Man Kin Wong, MBChB, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No